CLINICAL TRIAL: NCT03464123
Title: Brain Oxygenation During Cardiopulmonary Resuscitation - Observational Pilot Study
Brief Title: Brain Oxygenation During Cardiopulmonary Resuscitation
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Jouni Nurmi, MD, Consultant in Anaesthesia and Intensive Care Medicine, Helsinki University Central Hospital
Other Study IDs: 54/13/03/02/16
Record Dates: First submitted 2018-02-09; First posted 2018-03-13 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Cardiac Arrest, Out-Of-Hospital
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standard cardiopulmonary resuscitation — Standard Advanced Life Support based on guidelines 2015, including mechanical chest compression device

SUMMARY:
The study is aimed to assess (a) the incidence of hyperoxia at the point of return of spontaneous circulation (ROSC) and (b) the role of arterial blood oxygen partial pressure to brain oxygenation during out-of-hospital cardiac arrest. 80 adult patients will be recruited in a physician staffed helicopter emergency medical services. Brain regional oxygen saturation and invasive blood pressure are monitored until hospital admission and arterial blood gases are analyzed immediately when the unit arrives to the patient and again at the time of ROSC.

ELIGIBILITY:
Inclusion Criteria:

* out-of-hospital cardiac arrest of presumed cardiac origin
* resuscitation will be continued at least 5 minutes (if return of spontaneous circulation not achieved earlier) after arrival of physician team

Exclusion Criteria:

* do-not-attempt-resuscitation (DNAR) order or withdrawal of treatment by prehospital critical care physician
* return of spontaneous circulation achieved before physician-led critical team arrives
* external cause for cardiac arrest (e.g. trauma, suffocation)
* workload too high or environment too dangerous to perform study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients met in cardiac arrest by the physician-led prehospital critical care team are to be screened and recruited based the eligibility criteria. The patients include patients in all primary rhythms.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Arterial oxygen partial pressure | 5-60 minutes
  Arterial oxygen partial pressure at the time of return of spontaneous circulation (ROSC)

SECONDARY OUTCOMES:
Forehead regional oxygen saturation during resuscitation | 0-60 minutes
  Oxygen saturation measured using near-infrared spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Jouni Nurmi, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- FinnHEMS 10, Emergency Medicine and Services, Helsinki University Hospital, Vantaa, Finland

IPD SHARING:
Plan to Share IPD: No